CLINICAL TRIAL: NCT06880393
Title: A Study of BCMA CAR-T for Dynamic High-risk Patients With Multiple Myeloma
Brief Title: BCMA CAR-T for Dynamic High-risk Multiple Myeloma
Acronym: CAREMM-003
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024103
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA CAR-T (Experimental): Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA CAR+T cells/kg.
  Interventions: Biological: anti-BCMA-CAR-T

INTERVENTIONS:
Biological: anti-BCMA-CAR-T — Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2.0-4.0 x 10^6 anti-BCMA CAR+T cells/kg

SUMMARY:
This is a single-arm, open-label study to evaluate the efficacy and safety of BCMA CAR-T in dynamic high-risk patients with multiple myeloma

DETAILED DESCRIPTION:
The study is a prospective, single-arm, single-centre, phase II study designed to evaluate the efficacy and safety of BCMA CAR-T in dynamic high-risk patients with multiple myeloma. Patients received BCMA CAR-T cells infusion after standard FC lymphoma deletion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed and voluntarily sign the Informed Consent Form (ICF).
2. Age between 18 and 75 years (inclusive).
3. Have measurable disease meeting at least one of the following criteria: Serum M-protein ≥1 g/dL (>10 g/L) as detected by serum protein electrophoresis (SPEP), or quantifiable IgA or IgD levels for IgA or IgD-type myeloma; Urine M-protein ≥200 mg/24 hours; In cases where serum and urine M-protein do not meet the above thresholds, an abnormal free light chain (FLC) ratio (normal range: 0.26 to 1.65) and involved serum FLC ≥100 mg/L.
4. Have received only one line of standard anti-myeloma therapy, including: Induction therapy with at least one proteasome inhibitor, one immunomodulatory agent, and corticosteroids; Sequential autologous hematopoietic stem cell transplantation or consolidation therapy; Maintenance therapy based on either a proteasome inhibitor or an immunomodulatory agent.
5. Meet at least one of the following dynamic high-risk criteria: Early relapse: Disease progression or relapse within 18 months of starting first-line therapy, including progression or relapse within 12 months post-autologous hematopoietic stem cell transplantation; Primary refractory disease: Failure to achieve at least minimal response (MR) after four cycles of induction therapy; Relapse with new genetic abnormalities: Gain(1q), del(17p), or TP53 mutation.
6. Confirmed expression of the BCMA target antigen on MM cells by flow cytometry or bone marrow immunohistochemistry.

Exclusion Criteria:

1. Primary plasma cell leukemia.
2. Concurrent amyloidosis.
3. Involvement of the central nervous system (CNS).
4. Previous treatment with BCMA-targeted therapy or CAR-T cell therapy.
5. Disease progression or relapse within 3 months of autologous hematopoietic stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 2 year
  The incidence of treatment-emergent adverse events (TEAEs)
MRD-negative rate | within 3 months after BCMA CAR-T infusion
  achieving MRD-negative, as determined by NGS/NGF after consolidation treatment
Persistent MRD-negative rate | Up to 2 year
  Persistent MRD-negative rate more than 12 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first
Complete response rate (CRR) | within 3 month after the CAR-T cell transfusion
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No